CLINICAL TRIAL: NCT00273715
Title: A Comparative Randomized Efficacy Study of Sutures Versus Staples in Hip Surgical Procedures
Brief Title: Study of Sutures Versus Staples for Skin Closure After Surgical Procedures of Hip
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Kentucky (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-0715-F2L
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Surgery
Keywords: Comparative; Randomized; Suture; Staples, surgical; Skin; Surgical procedures, operative; Orthopedics; Joint, hip; Surgical procedures of Hip, Operative
MeSH Terms: interventions — Wound Closure Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Staples (No Intervention)
  Interventions: Procedure: Surgical wound closure techniques; Procedure: Surgical wound closure techniques (Comparator)

INTERVENTIONS:
Procedure: Surgical wound closure techniques — Subjects will be randomized to either receive sutures or staples during the surical procedure to close the incision
Procedure: Surgical wound closure techniques (Comparator) — Subjects will be randomized to either receive sutures or staples during the surical procedure to close the incision

SUMMARY:
Skin closure either by sutures or staples is required after any surgical procedure of the hip.

The purpose of this study is to compare the amount of drainage between patients who have had either staples or sutures placed for skin closure.

DETAILED DESCRIPTION:
Skin closure either by sutures or staples is required after any surgical procedure of the hip.

The purpose of this study is to compare the amount of drainage between patients who have had either staples or sutures placed for skin closure.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be 18 years of age or greater
* The patient must need an operative procedure of hip

Exclusion Criteria:

* Patients who are unable to undergo surgery.
* Patients who have a history of clotting or bleeding abnormalities.
* Patients who have arthroscopic hip surgery.
* Patients who have infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2005-12; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Amount of drainage from skin closure site | up to 5 days following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Selby, MD, Principal Investigator — University of Kentucky Department of Orthopaedic Surgery
Locations (1):
- University of Kentucky Chandler Medical Center, Lexington, Kentucky, United States